CLINICAL TRIAL: NCT06111560
Title: Exploring the Influence of Clinical Factors on the Prognosis of Papillary Renal Cell
Brief Title: Exploring the Influence of Clinical Factors on the Prognosis of Papillary Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zheng fufu, Professor,Phd,Md, Sun Yat-sen University
Other Study IDs: IIT-2023-282
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with tumor progression or recurrence: Patients enrolled in our retrospective study with tumor progression or recurrence
  Interventions: Other: We do not have any interventions. This study is based on obseravation.
- Patients without tumor progression or recurrence: Patients enrolled in our retrospective study without tumor progression or recurrence
  Interventions: Other: We do not have any interventions. This study is based on obseravation.

INTERVENTIONS:
Other: We do not have any interventions. This study is based on obseravation. — observational retrospective study without any interventions

SUMMARY:
Patients with renal cell carcinoma who were admitted to the First Affiliated Hospital of Sun Yat-sen University from February 1, 2021, to February 1, 2022, and met the following inclusion and exclusion criteria were collected. Clinical factors influencing the prognosis of enrolled patients were retrospectively analyzed, and a predictive system was established based on this.

(Inclusion criteria: pathology of the surgical specimen confirmed the diagnosis of pRCC,b: age 18 years or older, c: localized RCC underwent radical nephrectomy or partial nephrectomy in our center.

Exclusion criteria:a: lack of original CT images, b: patients with malignant tumors of other systems, c: patients who lost follow-up.)

ELIGIBILITY:
Inclusion Criteria:

a: pathology of the surgical specimen confirmed the diagnosis of pRCC,b: age 18 years or older, c: localized RCC underwent radical nephrectomy or partial nephrectomy in our center

Exclusion Criteria:

a: lack of original CT images, b: patients with malignant tumors of other systems, c: patients who lost follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the enrolled patients were Asian(we are a affiliated hospital of a university based in Mailand china ).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Tumor progression | 12 months
  medical imaging examinations showed tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Su, Bachelor, Principal Investigator — First affiliated hospital, Sun Yat-sen univeristy